CLINICAL TRIAL: NCT03025958
Title: Concurrent Nimotuzumab and Intensity-modulated Radiotherapy for Elderly Patients With Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Radiation Plus Concurrent Nimotuzumab in Elderly Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, Director of department, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2016-HN04
Record Dates: First submitted 2017-01-10; First posted 2017-01-20 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab; Radiation

STUDY DESIGN:
Intervention Model Description: Concomitant nimotuzumab was given weekly at a dose of 200 mg from one week before the start of IMRT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab (Experimental): Elderly patients with locoregionally advanced nasopharyngeal carcinoma were given an initial dose of nimotuzumab (200 mg) 7days before receiving concurrent radiotherapy, weekly nimotuzumab (200 mg/week).
  Interventions: Drug: Nimotuzumab; Radiation: Radiation

INTERVENTIONS:
Drug: Nimotuzumab — Concomitant nimotuzumab was given weekly at a dose of 200 mg from one week before the start of IMRT.
  Other Names: humanized anti-epidermal factor receptor monoclonal antibody h-R3
Radiation: Radiation — Briefly, the dose prescribed was 70.4 Gy, 70.4 Gy, 60.8 Gy, and 54.4 Gy in 32 fractions delivered over 6 weeks at the periphery of the planning target volume (PTV)nx+rn, PTVnd, PTV1, and PTV2, respectively, using the simultaneous integrated boost technique.

SUMMARY:
Radiation Plus Concurrent Nimotuzumab in Elderly Patients With Locoregionally Advanced Nasopharyngeal Carcinoma

DETAILED DESCRIPTION:
Elderly patients with locoregionally advanced nasopharyngeal carcinoma were given an initial dose of nimotuzumab (200 mg) 7days before receiving concurrent radiotherapy, weekly nimotuzumab (200 mg/week).

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated and histologically confirmed locoregionally advanced nasopharyngeal carcinoma

Exclusion Criteria:

* A history of another invasive cancer, prior RT to the head and neck area, prior cytotoxic chemotherapy or anti-EGFR therapy or the presence of any serious medical conditions, supposed to live less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate at 1 month after radiotherapy | 1 month after radiotherapy
  CR was defined as a complete lack of unequivocal soft tissue mass in the primary site and cervical lymph nodes with a short axis of less than 10 mm assessed by fiber-optic nasopharyngoscopy and MRI of the head and neck according to the Response Evaluation Criteria in Solid Tumors V.1.1 (RECIST V.1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No